CLINICAL TRIAL: NCT04625426
Title: Evaluate the Efficacy of Two Advanced Skin Treatment Regimens in Treating Incontinence-associated Dermatitis: Cluster Randomization Study
Brief Title: Evaluation of Skin Cleansers and Skin Protectants in Management of Incontinence-associated Dermatitis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Early termination due to COVID-19 pandemic led to inability to reach planned sample size
Sponsor: Tan Tock Seng Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SIG18037
Record Dates: First submitted 2020-10-06; First posted 2020-11-12 (Actual); Results first posted 2021-05-05 (Actual); Last update posted 2021-05-05 (Actual); Status verified 2021-05

CONDITIONS: Incontinence-associated Dermatitis

STUDY DESIGN:
Intervention Model Description: Cluster randomised trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 3M No-Rinse Cleanser and 3M Cavilon Advanced Skin Protectant (Experimental): Skin cleanser: 3M No-Rinse Cleanser. Skin protectant: 3M Cavilon Advanced Skin Protectant (liquid acrylic tetrapolymer skin protectant layer).
  The skin cleanser was used during every episode of incontinence and the protectant was applied every three days as recommended by the manufacturer.
  Interventions: Device: 3M Cavilon No-Rinse Skin Cleanser and 3M Cavilon Advanced Skin Protectant
- Conveen EasiCleanse and Conveen Critic Barrier (Experimental): Skin cleanser: Conveen EasiCleanse. Skin protectant: Conveen Critic Barrier (zinc oxide-based barrier cream). After each episode of incontinence, the skin cleanser was also first used to cleanse the skin, followed by application of the barrier cream, as per the barrier cream manufacturer's instructions.
  Interventions: Device: Conveen EasiCleanse and Conveen Critic Barrier
- Soap and water / Incontinence wipes and Conveen Critic Barrier (Active Comparator): Skin cleanser: Ordinary soap and water or incontinence wipes. Skin protectant: Conveen Critic Barrier (zinc oxide-based barrier cream). After each episode of incontinence, the skin was cleansed using soap and water or incontinence wipes, followed by application of the barrier cream.
  Interventions: Device: Standard cleansing and Conveen Critic Barrier

INTERVENTIONS:
Device: 3M Cavilon No-Rinse Skin Cleanser and 3M Cavilon Advanced Skin Protectant — Hypoallergenic no-rinse skin cleanser and liquid acrylic tetrapolymer skin protectant
  Arms: 3M No-Rinse Cleanser and 3M Cavilon Advanced Skin Protectant
Device: Conveen EasiCleanse and Conveen Critic Barrier — Hypoallergenic no-rinse skin cleanser and zinc-oxide barrier cream
  Arms: Conveen EasiCleanse and Conveen Critic Barrier
Device: Standard cleansing and Conveen Critic Barrier — Hospital's standard care for IAD management
  Arms: Soap and water / Incontinence wipes and Conveen Critic Barrier

SUMMARY:
The aim of this study is to evaluate the efficacy of two different skin care regimens (3M Cavilon Advanced Skin Protectant with 3M No-Rinse Cleanser and Coloplast Conveen Critic Barrier with Easi-Cleanser) against standard care (Skin wipes and Conveen Critic Barrier) in the management of Incontinence-Associated Dermatitis (IAD) in hospitalised patients

DETAILED DESCRIPTION:
The aim of this study is to evaluate the efficacy of two different skin care regimens (3M Cavilon Advanced Skin Protectant with 3M No-Rinse Cleanser and Coloplast Conveen Critic Barrier with Easi-Cleanser) against standard care (Skin wipes and Conveen Critic Barrier) in the management of Incontinence-Associated Dermatitis (IAD) in hospitalised patients.

To date, there is no conclusive evidence on the "best treatment" for patients presenting with IAD. This has led to current clinical practices tend to select IAD products based on its cost and availability, which can be heavily influenced by marketing and commercialisation efforts.

This study allows investigation of the effectiveness of IAD products to ensure the provision of optimal care.

ELIGIBILITY:
Inclusion Criteria:

* Aged 21 years and above at point of recruitment
* Diagnosed with IAD
* At regular risk of exposure to urine and faeces over their hospitalization

Exclusion Criteria:

* Having a known allergy to the treatment products
* Haemodynamically unstable at point of assessment for study
* Unable to tolerate lateral positioning for skin cleansing and treatment application
* Pregnancy
* Having an existing skin disease at point of study that might lead to inaccurate IAD assessment, such as herpes or scabies.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2019-04-29 (Actual); Primary Completion 2020-01-20 (Actual); Study Completion 2020-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ee Yuee Chan, Study Director — Tan Tock Seng Hospital; Cheng Cheng Goh, Principal Investigator — Tan Tock Seng Hospital
Locations (1):
- Tan Tock Seng Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
No plans to share IPD to other researchers.

REFERENCES:
- [Background] Beeckman D, Van Damme N, Schoonhoven L, Van Lancker A, Kottner J, Beele H, Gray M, Woodward S, Fader M, Van den Bussche K, Van Hecke A, De Meyer D, Verhaeghe S. Interventions for preventing and treating incontinence-associated dermatitis in adults. Cochrane Database Syst Rev. 2016 Nov 10;11(11):CD011627. doi: 10.1002/14651858.CD011627.pub2. PMID 27841440
- [Background] Van Tiggelen H, LeBlanc K, Campbell K, Woo K, Baranoski S, Chang YY, Dunk AM, Gloeckner M, Hevia H, Holloway S, Idensohn P, Karadag A, Koren E, Kottner J, Langemo D, Ousey K, Pokorna A, Romanelli M, Santos VLCG, Smet S, Tariq G, Van den Bussche K, Van Hecke A, Verhaeghe S, Vuagnat H, Williams A, Beeckman D. Standardizing the classification of skin tears: validity and reliability testing of the International Skin Tear Advisory Panel Classification System in 44 countries. Br J Dermatol. 2020 Jul;183(1):146-154. doi: 10.1111/bjd.18604. Epub 2019 Nov 28. PMID 31605618
- [Background] Beele H, Smet S, Van Damme N, Beeckman D. Incontinence-Associated Dermatitis: Pathogenesis, Contributing Factors, Prevention and Management Options. Drugs Aging. 2018 Jan;35(1):1-10. doi: 10.1007/s40266-017-0507-1. PMID 29243033

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 2 participants initially recruited were found to be not eligible before being assigned to an arm, leading to them being dropped from the study before assignation.
Groups:
- 3M No-Rinse Cleanser and 3M Cavilon Advanced Skin Protectant: Skin cleanser: 3M No-Rinse Cleanser. Skin protectant: 3M Cavilon Advanced Skin Protectant (liquid acrylic tetrapolymer skin protectant layer).
  The skin cleanser was used during every episode of incontinence and the protectant was applied every three days as recommended by the manufacturer.
  3M Cavilon No-Rinse Skin Cleanser and 3M Cavilon Advanced Skin Protectant: Hypoallergenic no-rinse skin cleanser and liquid acrylic tetrapolymer skin protectant
Period: Overall Study
Arm/Group | 3M No-Rinse Cleanser and 3M Cavilon Advanced Skin Protectant | Conveen EasiCleanse and Conveen Critic Barrier | Soap and Water / Incontinence Wipes and Conveen Critic Barrier
Started | 23 | 37 | 24
Completed | 9 | 12 | 12
Not Completed | 14 | 25 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 3M No-Rinse Cleanser and 3M Cavilon Advanced Skin Protectant | Conveen EasiCleanse and Conveen Critic Barrier | Soap and Water / Incontinence Wipes and Conveen Critic Barrier | Total
Number analyzed (Participants) | 23 | 37 | 24 | 84
Age, Continuous [Mean (Standard Deviation); unit: years] | 77.2 (10.6) | 80.2 (9.56) | 80.7 (8.03) | 79.51 (9.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 20 | 12 | 46
  Male | 9 | 17 | 12 | 38
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Chinese | 22 | 35 | 22 | 79
  Malay | 0 | 2 | 0 | 2
  Indian | 1 | 0 | 2 | 3
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 20.3 (3.81) | 21.0 (5.19) | 20.4 (3.42) | 20.6 (4.18)
Type of incontinence [Number; unit: participants]
  Urinary incontinence | 17 | 24 | 21 | 62
  Faecal incontinence | 22 | 37 | 24 | 83
  Dual incontinence | 16 | 24 | 21 | 61
Faecal frequency [Mean (Standard Deviation); unit: episodes/day] | 3.25 (1.65) | 3.52 (2.01) | 3.43 (2.31) | 3.43 (2.01)
Presence of indwelling urinary catheter [Count of Participants; unit: Participants] | 7 | 12 | 3 | 22
Stool consistency [Count of Participants; unit: Participants] — Stool consistency measured using Bristol Stool Chart. The chart grades stool by 7 types Types 3 and 4 are ideal, reflecting smooth,easy-to-pass stool Types 1 and 2 are not ideal as they indicate diarrhoea Types 5, 6 and 7 are not ideal as they indicate diarrhoea Type 1: Separate hard lumps, hard to pass Type 2: Separate hard lumps, hard to pass Type 3, Type 4: Ideal stool consistency, smooth Type 5: Soft blobs with clear-cut edges Type 6: Mushy, fluffy stool Type 7: Watery, entirely liquid
  Participants
    Type 4 (Best Outcome) | 0 | 2 | 3 | 5
    Type 5 (Second-best) | 4 | 8 | 4 | 16
    Type 6 (Third-best outcome) | 6 | 12 | 8 | 26
    Type 7 (Worst outcome) | 6 | 9 | 6 | 21
    Missing | 7 | 6 | 3 | 16

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced IAD Healing
Description: Total number of participants who experienced IAD healing
Time Frame: Up to seven days from initiation of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | 3M No-Rinse Cleanser and 3M Cavilon Advanced Skin Protectant | Conveen EasiCleanse and Conveen Critic Barrier | Soap and Water / Incontinence Wipes and Conveen Critic Barrier
Number analyzed (Participants) | 23 | 37 | 24
Participants
  Healed | 8 | 12 | 5
  Censored | 15 | 25 | 19

2. Primary Outcome: Proportion of Participants With IAD Healing
Description: Percentage of participants who experienced IAD healing
Time Frame: Up to seven days from initiation of treatment
Measure: Number; unit: percentage of participants
Arm/Group | 3M No-Rinse Cleanser and 3M Cavilon Advanced Skin Protectant | Conveen EasiCleanse and Conveen Critic Barrier | Soap and Water / Incontinence Wipes and Conveen Critic Barrier
Number analyzed (Participants) | 23 | 37 | 24
percentage of participants | 35 | 32 | 21

3. Secondary Outcome: Number of Participants Who Developed Skin Loss
Description: Examination of the development of skin loss using the Ghent Global IAD Categorisation tool (GLOBIAD).
  Binary scoring, 1 and 2. Higher value (2) indicates worse outcome (Development of skin loss)
Time Frame: Up to three days from initiation of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | 3M No-Rinse Cleanser and 3M Cavilon Advanced Skin Protectant | Conveen EasiCleanse and Conveen Critic Barrier | Soap and Water / Incontinence Wipes and Conveen Critic Barrier
Number analyzed (Participants) | 23 | 37 | 24
Participants | 0 | 5 | 3

ADVERSE EVENTS:
Time Frame: Adverse data not collected over study period. This is because the interventions were assessed to have minimal risk of harm on participants.
Description: All-Cause Mortality, Serious and Other [Not Including Serious] Adverse Events were not monitored/assessed as interventions were assessed to have minimal risk of harm on participants.
Arm/Group | 3M No-Rinse Cleanser and 3M Cavilon Advanced Skin Protectant | Conveen EasiCleanse and Conveen Critic Barrier | Soap and Water / Incontinence Wipes and Conveen Critic Barrier
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Early termination due to COVID-19 pandemic led to inability to reach planned sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-05): https://cdn.clinicaltrials.gov/large-docs/26/NCT04625426/Prot_SAP_000.pdf